CLINICAL TRIAL: NCT07038746
Title: A Phase 1b, Open-Label, Exploratory Study Evaluating the Effects of Inhaled Epinephrine in Individuals Experiencing Systemic Allergic Reactions During Allergy Testing, Immunotherapy or Oral Challenges
Brief Title: Effects of Inhaled Epinephrine on Systemic Allergic Reactions During Allergy Testing, Immunotherapy or Oral Challenges
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. George Luciuk (Other)
Responsible Party: Sponsor-Investigator, Dr. George Luciuk, President, Chief Medical Officer, Kokua Pharma Inc.
Organization: Kokua Pharma Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHL-102
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hypersensitivity; Anaphylaxis
Keywords: Immunotherapy; Epinephrine; Upper airway laryngeal edema; Upper airway pharyngeal edema; Hypersensitivity; Hypersensitivity, immediate; Anaphylaxis; Vasoconstrictor agents; Adrenergic alpha-Agonists; Adrenergic beta-Agonists; Bronchodilator agents
MeSH Terms: conditions — Hypersensitivity; Anaphylaxis; Hypersensitivity, Immediate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Inhaled Epinephrine (Experimental): The first inhalation will be administered as soon as possible (i.e., within approximately 30 seconds) following identification of a SAR Grade 2 or higher and confirmation of enrollment by the Principal Investigator. The second inhalation will be administered approximately 10 seconds later, and the subject will be observed for approximately 2 minutes for signs of symptom resolution.
  Inhalations will continue in this manner until either:
  1. resolution of systemic symptoms (defined as a reduction in SAR Grade to ≤1), or
  2. if maximum number of inhalations (8 inhalations) has not been reached, complete resolution of systemic symptoms (defined as reduction in SAR Grade to 0) without exceeding maximum 8 inhalations, or
  3. administration of intra-muscular epinephrine, whichever occurs earlier.
  If a recurrence of symptoms is observed, administration may continue until a maximum of 8 inhalations is reached.
  Interventions: Drug: Inhaled Epinephrine

INTERVENTIONS:
Drug: Inhaled Epinephrine — 0.125 mg per inhalation.
  The maximum proposed dose to be administered is 1.0 mg (consisting of 8 inhalations of 0.125 mg over 6 minutes).

SUMMARY:
The goal of this exploratory study is to evaluate the effects of inhaled epinephrine in subjects, who may not be eligible for the GHL-101 trial, and who are experiencing systemic allergic reaction (SAR) that occur following allergy testing, subcutaneous immunotherapy (SCIT), oral challenges (with food and/or drug) or oral immunotherapy (OIT).

DETAILED DESCRIPTION:
This is a Phase 1b, multi-center, open label exploratory study evaluating the effects of inhaled epinephrine in patients who are undergoing planned allergy testing, SCIT, oral challenges (with food and/or drug), or OIT and are not eligible for the GHL-101 study. This study will enroll and dose up to 100 patients.

The maximum duration of subject participation is approximately 1 week.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged ≥ 12 years with known or suspected allergen sensitivity who can also have a clinical history of immunoglobulin E (IgE)-mediated allergy, including a documented sensitivity to allergens (i.e., positive skin prick test, or positive in vitro serum IgE).
2. Have undergone either a) allergy testing for suspected sensitivity/allergy, b) future oral challenge (food and/or drug) or future OIT to treat existing allergies or c) SCIT AND experienced a SAR Grade 2 or higher, following allergy testing, SCIT, or oral challenges (food and/or drug) for future OIT, and deemed eligible for enrollment by the Principal Investigator.
3. For females of child-bearing potential, not pregnant or lactating, willing to use an acceptable contraception* method between Screening and End-of-Study Visits.

Exclusion Criteria:

1. Known reaction or sensitivity to epinephrine or any of the ingredients of inhaled epinephrine.
2. Known history or presence of clinically disease/condition that could confound the results of the study or place the subject at undue or additional risk per the judgment of the Investigator.
3. Abnormal vital signs at screening (i.e., systolic blood pressure: < 90 or >140 mmHg, diastolic blood pressure: < 40 or > 90 mmHg or, heart rate: < 45 or > 100 bpm), respiration rate < 8 or > 20 resp./min.
4. Females who are pregnant, plan to become pregnant or lactating.
5. Participation in another clinical study involving an investigational drug within 30 days prior to screening, an investigational biologic within 60 days prior to screening, or current/planned participation in another interventional study during this study.
6. Previous treatment in this study.
7. Any other reason that, in the opinion of the Investigator, is likely to unfavorably alter subject risk-benefit, confound results, or make it difficult for the subject to fully comply with study requirements.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of systemic symptoms | From first dose administration to 60 minutes following first dose administration
  Defined as a reduction in systemic allergic reaction (SAR) Grade to ≤ 1. Grade 0 is considered the absence of any symptoms and per World Allergy Organisation's Grading System for Systemic Allergic Reactions, Grade 1 is least severe and Grade 5 is most severe.
Time to complete resolution of systemic symptoms | From first dose administration to 60 minutes following first dose administration
  Defined as a reduction in systemic allergic reaction (SAR) Grade to 0. Grade 0 is considered the absence of any symptoms and per World Allergy Organisation's Grading System for Systemic Allergic Reactions, Grade 1 is least severe and Grade 5 is most severe.

CONTACTS AND LOCATIONS:
Overall Officials: George H. Luciuk, MD, Principal Investigator — Kokua Pharma Inc.
Locations (1):
- Kokua Pharma Inc., Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately after publication, and for a period of 5 years.
Access Criteria: Any purpose. URL to be added.